CLINICAL TRIAL: NCT01662856
Title: A Prospective, Single-blind, Randomized, Phase III Study to Evaluate the Safety and Efficacy of Fibrin Sealant Grifols (FS Grifols) as an Adjunct to Hemostasis During Peripheral Vascular Surgery
Brief Title: Safety and Efficacy Study of Fibrin Sealant Grifols as an Adjunct to Hemostasis During Peripheral Vascular Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Grifols, S.A. (Industry)
Responsible Party: Sponsor
Organization: Grifols Biologicals, LLC (Industry)
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: IG1101
Record Dates: First submitted 2012-08-07; First posted 2012-08-10 (Estimated); Results first posted 2017-04-06 (Actual); Last update posted 2017-04-06 (Actual); Status verified 2017-02

CONDITIONS: Vascular Surgical Bleeding
Keywords: Vascular Surgery; Fibrin Sealant; Polytetrafluoroethylene (PTFE) grafts

ARMS (2):
- Fibrin Sealant Grifols (Experimental): Fibrin Sealant Grifols consisting of 3 mL fibrinogen and 3 mL thrombin in separate syringes assembled on a syringe holder (6 mL of solution in total).
  Interventions: Biological: Fibrin Sealant Grifols
- Manual Compression (Active Comparator): Direct manual compression of target bleeding site with gauze/laparotomy pads.
  Interventions: Procedure: Manual Compression

INTERVENTIONS:
Biological: Fibrin Sealant Grifols — Combination of 3 mL fibrinogen and 3 mL thrombin in separate syringes assembled on a syringe holder (6 mL of solution in total).
  Arms: Fibrin Sealant Grifols
Procedure: Manual Compression — Direct manual compression of target bleeding site with gauze/laparotomy pads.
  Arms: Manual Compression

SUMMARY:
The purpose of this study is to demonstrate that the application of Fibrin Sealant Grifols provides a measurable benefit when compared to hemostasis achieved through conventional surgical technique (suture) and by standard hemostatic action, such as mechanical pressure through manual compression. This study has a Preliminary Part (I) in which all subjects are treated with Fibrin Sealant Grifols and a Primary Part (II) in which subjects are randomized in a 2:1 ratio to either Fibrin Sealant Grifols or manual compression.

ELIGIBILITY:
Inclusion Criteria:

* Hemoglobin (Hgb) ≥ 8.0 g/dL at Baseline (within 24 hours prior to surgical procedure).
* Require elective (non-emergency), primary, open (non-laparoscopic; non-endovascular) peripheral vascular surgery.
* Require one of the following peripheral vascular procedures involving proximal end-to-side arterial anastomosis utilizing coated or uncoated Polytetrafluoroethylene grafts: a) Femoral-femoral bypass grafting, b) Femoral-popliteal bypass grafting, c) Femoral-distal bypass grafting, d) Ilio-iliac bypass grafting, e) Ilio-femoral bypass grafting, f) Ilio-popliteal bypass grafting, g) Aorto-iliac bypass grafting, h) Aorto-femoral bypass grafting, i)Axillo-femoral bypass grafting, and j) Upper extremity vascular access for hemodialysis.
* A target bleeding site can be identified.
* Target bleeding site has moderate arterial bleeding.

Exclusion Criteria:

* Undergoing a re-operative procedure.
* Undergoing other vascular procedures during the same surgical session (stenting and/or endarterectomy of the same artery are allowed).
* Have an infection in the anatomic surgical area.
* Have a history of severe (e.g. anaphylactic) reactions to blood or to any blood-derived product.
* Have previous known sensitivity to any Fibrin Sealant Grifols, heparin, or protamine component.
* Females who are pregnant or nursing a child at Baseline (within 24 hours prior to surgical procedure).
* Have undergone a therapeutic surgical procedure within 30 days from the screening visit.
* Target bleeding site cannot be identified.
* Target bleeding site has mild or severe arterial bleeding.
* Occurrence of major intraoperative complications that require resuscitation or deviation from the planned surgical procedure.
* Intraoperative change in planned surgical procedure, which results in subject no longer meeting preoperative inclusion and/or exclusion criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2012-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (38):
- United States (27):
  - 407, Florence, Alabama
  - 125, Palo Alto, California
  - 119, San Diego, California
  - 149, Jacksonville, Florida
  - 148, Jacksonville, Florida
  - 137, Tampa, Florida
  - 140, Atlanta, Georgia
  - 114, Iowa City, Iowa
  - 110, Lexington, Kentucky
  - 146, Baton Rouge, Louisiana
  - 132, New Orleans, Louisiana
  - 129, Baltimore, Maryland
  - 135, Bethesda, Maryland
  - 102, Boston, Massachusetts
  - 406, Manhasset, New York
  - 113, Stony Brook, New York
  - 142, The Bronx, New York
  - 409, Dayton, Ohio
  - 104, Toledo, Ohio
  - 100, 128, Pittsburgh, Pennsylvania
  - 115, West Reading, Pennsylvania
  - 147, Fort Worth, Texas
  - 402, Houston, Texas
  - 139, Salt Lake City, Utah
  - 103, Seattle, Washington
  - 138, Tacoma, Washington
  - 111, Madison, Wisconsin
- Hungary (3):
  - 501, Miskolc
  - 500, Pécs
  - 502, Veszprém
- Russia (5):
  - 540, Novosibirsk
  - 542, Rostov-on-Don
  - 541, Saint Petersburg
  - 543, Saint Petersburg
  - 544, Saint Petersburg
- Serbia (3):
  - 523, Belgrade
  - 521, Belgrade
  - 522,524, Novi Sad

REFERENCES:
- [Derived] Ma GW, Kucey A, Tyagi SC, Papia G, Kucey DS, Varcoe RL, Forbes T, Neville R, Dueck AD, Kayssi A. The role of sealants for achieving anastomotic hemostasis in vascular surgery. Cochrane Database Syst Rev. 2024 May 2;5(5):CD013421. doi: 10.1002/14651858.CD013421.pub2. PMID 38695613

RESULTS

PARTICIPANT FLOW:
Groups:
- Fibrin Sealant Grifols: Fibrin Sealant Grifols consisting of 3 mL fibrinogen and 3 mL thrombin in separate syringes assembled on a syringe holder (6 mL of solution in total), applied topically to target bleeding site.
Period: Part I + Part II (Overall Study)
Arm/Group | Fibrin Sealant Grifols | Manual Compression
Started | 168 | 57
Completed Study up to Week 6 | 164 | 56
Completed | 152 (Completed Virology follow-up visit at Month 3 or Month 6) | 55 (Completed Virology follow-up visit at Month 3 or Month 6)
Not Completed | 16 | 2
Period: Primary Part II
Arm/Group | Fibrin Sealant Grifols | Manual Compression
Started | 109 | 57
Completed Study up to Week 6 | 106 | 56
Completed | 99 (Completed Virology follow-up visit at Month 3 or Month 6) | 55 (Completed Virology follow-up visit at Month 3 or Month 6)
Not Completed | 10 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fibrin Sealant Grifols | Manual Compression | Total
Number analyzed (Participants) | 168 | 57 | 225
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.65 (9.036) | 62.04 (10.734) | 63.24 (9.496)
Age, Customized [Number; unit: participants]
  Between 18 and 64 years | 90 | 32 | 122
  >=65 years | 78 | 25 | 103
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 26 | 77
  Male | 117 | 31 | 148
Region of Enrollment [Number; unit: participants]
  Russian Federation | 18 | 3 | 21
  Hungary | 49 | 23 | 72
  United States | 69 | 16 | 85
  Serbia | 32 | 15 | 47

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Achieving Hemostasis by Four Minutes After Treatment Start
Description: Subjects achieving hemostasis at the target bleeding site by 4 minutes following the start of treatment without the occurrence of re-bleeding until the completion of surgical closure.
Time Frame: From start of treatment until 4 minutes after treatment start
Population: Efficacy analysis was performed on subjects in the Primary Part (II) of the study
Measure: Number; unit: Percent of subjects achieving hemostasis
Arm/Group | Fibrin Sealant Grifols | Manual Compression
Number analyzed (Participants) | 109 | 57
Percent of subjects achieving hemostasis | 76.1 | 22.8

2. Secondary Outcome: Time to Hemostasis (TTH)
Description: Time in minutes for achievement of hemostasis at the target bleeding site measured from the start of treatment until 10 minutes after treatment start.
  In the Fibrin Sealant Grifols treatment group, the median TTH was calculated based on the estimated survival function S(t), and it is the smallest time at which S(t) is at or below 50%. The 95% CI for the median TTH, on the other hand, was calculated based on the CI for the survival function S(t). The 95% CI for the median TTH was the set of all time points for which the 95% CI of the survival function contains 0.5 (since median is the 50% percentile). Sometimes, the confidence limits for the median cannot be estimated. In our case, the hemostasis was assessed on a discrete scale, and it happened that for all the time points assessed none of the 95% CI of the survival function S(t) contained 0.5. As a result, neither the lower nor the upper limit could be estimated.
  All calculations were performed using SAS PROC LIFETEST
Time Frame: From start of treatment until 10 minutes after treatment start
Population: Efficacy analysis was performed on subjects in the Primary Part (II) of the study
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Fibrin Sealant Grifols | Manual Compression
Number analyzed (Participants) | 109 | 57
minutes | 4.0 [NA to NA] — Neither the lower nor upper 95% CI limit for median TTH could be estimated; for all time points with hemostatic assessment, none of the 95% CIs of the S(t) contained 0.5 (corresponding to the 50th percentile, ie, median). See Measure Description. | NA [10.00 to NA] — Median TTH could not be estimated precisely; most subjects did not achieve hemostasis by 10 minutes after start of treatment and were considered censored. Lower limit of the 95% CI was 10 minutes, it was deduced that the median TTH was ≥10 minutes.

3. Secondary Outcome: Cumulative Proportion of Subjects Having Achieved Hemostasis at the Target Bleeding Site by Specified Time Points
Description: Cumulative proportion of subjects having achieved hemostasis by each of the following time points:
  * At 5 minutes following start of study treatment
  * At 7 minutes following start of study treatment
  * At 10 minutes following start of study treatment
Time Frame: From start of treatment until 10 minutes after treatment start
Population: Efficacy analysis was performed on subjects in the Primary Part (II) of the study
Measure: Number; unit: Percent of subjects achieving hemostasis
Arm/Group | Fibrin Sealant Grifols | Manual Compression
Number analyzed (Participants) | 109 | 57
Percent of subjects achieving hemostasis
  Hemostasis by 5 minutes | 80.7 | 28.1
  Hemostasis by 7 minutes | 84.4 | 35.1
  Hemostasis by 10 minutes | 88.1 | 45.6

4. Secondary Outcome: Prevalence of Treatment Failures
Description: Protocol-defined bleeding at the target bleeding site after the start of treatment or the use of alternative hemostatic treatments (with exception of reversal of heparin) or maneuvers at the target bleeding site after the start of treatment.
Time Frame: From start of treatment until 10 minutes after treatment start
Population: Efficacy analysis was performed on subjects in the Primary Part (II) of the study
Measure: Number; unit: percent of subjects
Arm/Group | Fibrin Sealant Grifols | Manual Compression
Number analyzed (Participants) | 109 | 57
percent of subjects | 23.9 | 77.2

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time informed consent was obtained through the Post-Operative Week 6 (±4 days) Visit
Arm/Group | Fibrin Sealant Grifols | Manual Compression
Serious Adverse Events (participants affected / at risk) | 34/168 | 11/57
Other Adverse Events (participants affected / at risk) | 132/168 | 41/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fibrin Sealant Grifols (N=168) | Manual Compression (N=57)
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 2 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Diabetic gastroparesis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Death (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 0
Cellulitis (Infections and infestations) | 2 | 0
Endocarditis (Infections and infestations) | 1 | 0
Gangrene (Infections and infestations) | 1 | 2
Graft infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 0
Postoperative wound infection (Infections and infestations) | 3 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 2 | 0
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Reocclusion (Injury, poisoning and procedural complications) | 2 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 | 0
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 1 | 2
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 0
Parvovirus B19 test positive (Investigations) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carotid sinus syndrome (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0
Lymphorrhoea (Vascular disorders) | 1 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fibrin Sealant Grifols (N=168) | Manual Compression (N=57)
Anaemia (Blood and lymphatic system disorders) | 10 | 2
Constipation (Gastrointestinal disorders) | 7 | 4
Nausea (Gastrointestinal disorders) | 10 | 2
Vomiting (Gastrointestinal disorders) | 4 | 3
Oedema peripheral (General disorders) | 13 | 1
Pyrexia (General disorders) | 19 | 6
Anaemia postoperative (Injury, poisoning and procedural complications) | 9 | 2
Procedural pain (Injury, poisoning and procedural complications) | 58 | 21
Body temperature increased (Investigations) | 10 | 4
Hypotension (Vascular disorders) | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site may publish results from the Study, after providing Sponsor thirty days' notice prior to submitting a manuscript or other materials related to the Study to any outside party. At Sponsors' request, Site will remove any Confidential Information (other than Study results), and Site will upon Sponsors' request, delay publication or presentation for a period of up to one hundred twenty days to allow Sponsor to protect its interests in any Sponsor Inventions.